CLINICAL TRIAL: NCT00054067
Title: Treatment of Patients With Stage IB2 Carcinoma of the Cervix: A Randomized Comparison of Radical Hysterectomy and Tailored Chemo-Radiation Versus Primary Chemo-Radiation
Brief Title: Chemotherapy and Radiation Therapy With or Without Surgery in Treating Patients With Stage I Cancer of the Cervix
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: GOG Foundation (Network)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000269821; GOG-0201
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2013-04

CONDITIONS: Cervical Cancer
Keywords: cervical adenocarcinoma; cervical adenosquamous cell carcinoma; cervical squamous cell carcinoma; stage IB cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Cisplatin; Chemotherapy, Adjuvant; Brachytherapy; Radiotherapy

INTERVENTIONS:
Drug: cisplatin
Procedure: adjuvant therapy
Procedure: conventional surgery
Radiation: brachytherapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known which regimen of radiation therapy combined with chemotherapy, with or without surgery, is more effective in treating early cancer of the cervix.

PURPOSE: Randomized phase III trial to compare the effectiveness of surgery followed by different regimens of radiation therapy and chemotherapy with that of chemotherapy and radiation therapy alone in treating patients who have stage I cancer of the cervix.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare progression-free survival and survival of patients with stage IB2 carcinoma of the cervix after radical hysterectomy with tailored chemoradiotherapy vs primary chemoradiotherapy.
* Compare the toxicity of these regimens in these patients.
* Compare the health-related quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: (Surgery followed by chemoradiotherapy): Patients undergo exploratory laparotomy followed by radical hysterectomy and bilateral pelvic and para-aortic lymphadenectomy. Depending on the findings at surgery, the radical hysterectomy and lymphadenectomy are either completed or aborted.

  * Aborted hysterectomy: Patients with aborted hysterectomy are assigned to 1 of 3 groups, depending on the findings at surgery.

    * Group 1: Within 4 weeks of surgery, patients undergo pelvic radiotherapy 5 times weekly for 4-6 weeks and intracavitary irradiation during or after external radiotherapy. Patients also receive concurrent cisplatin IV over 1 hour once weekly for a total of 5-6 doses.
    * Group 2: Patients receive radiotherapy and cisplatin as in group 1 with additional extended field radiotherapy.
    * Group 3: Patients receive further treatment at the discretion of the investigator.
  * Completed hysterectomy: Patients completing the radical hysterectomy are assigned to 1 of 3 groups, depending on the findings at surgery.

    * Group A: Patients receive treatment as in group 1 above without intracavity irradiation.
    * Group B: Patients receive treatment as in group 2 above without intracavity irradiation.
    * Group C: Patients receive no further treatment.
* Arm II (Primary chemoradiotherapy): Patients undergo pelvic radiotherapy 5 times weekly for 4-6 weeks and intracavity irradiation during or after external radiotherapy. Patients also receive concurrent cisplatin IV over 1 hour once weekly for a total of 6 doses.

Quality of life is assessed at baseline, during week 5 of therapy, and then at 3, 6, and 12 months.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 740 patients (370 per treatment arm) will be accrued for this study within 7.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage IB2 invasive carcinoma of the uterine cervix of one of the following types:

  * Squamous cell carcinoma
  * Adenocarcinoma
  * Adenosquamous carcinoma
* Primary, previously untreated disease
* Exophytic cervical lesions greater than 4 cm in diameter OR
* Cervical expansion to greater than 4 cm in diameter, presumed to be the result of principal involvement with cancer
* No evidence of extrauterine disease other than pelvic lymph node involvement (by clinical and radiographic examinations)
* No para-aortic lymph nodal disease (suspected on CT scan, MRI, positron-emission tomography, or lymphangiogram) unless nodes are confirmed to be pathologically negative (by CT-guided biopsy or extraperitoneal lymph node dissection)
* Eligible for radical hysterectomy and lymph node dissection

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* GOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than 1.5 times normal
* SGOT no greater than 3 times normal
* Alkaline phosphatase no greater than 3 times normal

Renal

* Creatinine no greater than 2.0 mg/dL
* No renal abnormalities requiring modification of radiation fields

Gastrointestinal

* No gastrointestinal bleeding
* No intestinal obstruction

Other

* Not pregnant
* Negative pregnancy test
* No septicemia or severe infection
* No other invasive malignancy with any evidence of disease within the past 5 years except nonmelanoma skin cancer
* No circumstances that would preclude study completion or required follow-up

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy

Surgery

* See Disease Characteristics
* No prior hysterectomy (total or subtotal)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-02; Primary Completion 2005-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: D. Scott McMeekin, MD, Study Chair — Oklahoma University Cancer Institute
Locations (50):
- United States (49):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - CCOP - Western Regional, Arizona, Phoenix, Arizona
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Women's Cancer Center at Community Hospital of Los Gatos, Los Gatos, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Cancer Center, Orange, California
  - Yale Comprehensive Cancer Center, New Haven, Connecticut
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Cooper University Hospital, Camden, New Jersey
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Long Island Cancer Center at Stony Brook University Hospital, Stony Brook, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Abramson Cancer Center at University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Magee-Womens Hospital, Pittsburgh, Pennsylvania
  - Southeast Gynecologic Oncology Associates, Knoxville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Vanderbilt Medical Center, Nashville, Tennessee
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Fletcher Allen Health Care - Medical Center Campus, Burlington, Vermont
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
- Kagoshima City Hospital, Kagoshima, Japan